CLINICAL TRIAL: NCT03838601
Title: Role of Microbiome as a Biomarkers in Locoregionally-Advanced Oropharyngeal Squamous Cell Carcinoma 2 (ROMA LA-OPSCC-2)
Brief Title: Role of Microbiome as a Biomarkers in Locoregionally-Advanced Oropharyngeal Squamous Cell Carcinoma 2
Acronym: ROMA LA-OPSCC2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: NuBiyota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROMA LA-OPSCC-002
Record Dates: First submitted 2019-02-05; First posted 2019-02-12 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MET-4 (Experimental): Subjects diagnosed with Locoregionally-Advanced Oropharyngeal Squamous Cell Carcinoma (LA-OPSCC) will receive treatment with MET-4 in addition to standard of care CRT. MET-4 is administered orally as an initial daily loading dose over 2 days followed by a daily maintenance dose of MET-4 and will be administered until week 4 of CRT or unacceptable toxicity whichever occurs earlier and in the absence of criteria to discontinue MET-4.
  Interventions: Drug: MET-4

INTERVENTIONS:
Drug: MET-4 — Microbial Ecosystem Therapeutics (MET) is a new treatment approach developed as an alternative to fecal transplantation. Unlike donor stool used in fecal transplants, which are incompletely characterised complex communities of microbes and associated metabolites and fecal material, MET consists of a defined mixture of pure live cultures of intestinal bacteria isolated from a stool sample of a healthy donor.

SUMMARY:
This is a single-centre feasibility study designed to assess the safety, tolerability and engraftment of MET-4 bacterial strains when given in combination with chemoradiotherapy (CRT). The study will involve a prospective cohort of 30 patients diagnosed with Locoregionally-Advanced Oropharyngeal Squamous Cell Carcinoma (LA-OPSCC) to be treated with CRT as per standard of care at Princess Margaret Cancer Centre. All patients enrolled will receive MET-4 in addition to standard CRT. MET-4 is administered orally as an initial daily loading dose over 2 days followed by a daily maintenance dose of MET-4 and will be administered until week 4 of CRT or unacceptable toxicity whichever occurs earlier and in the absence of criteria to discontinue MET-4. This protocol does not determine eligibility to receive treatment with concurrent CRT. It is anticipated that patient accrual will be completed within 12 months.

DETAILED DESCRIPTION:
Past findings suggest oral microbiome might be used to predict recurrence and response to therapies, as past studies have shown surgery, radiotherapy and chemotherapy alter the microbiome, which in turn modulates treatment effectiveness/toxicity.

Microbial Ecosystem Therapeutics (MET) is a new treatment approach developed as an alternative to fecal transplantation. MET consists of a mixture of pure live cultures of intestinal bacteria isolated from stool of a healthy donor. MET-1 administered by colonoscopy was successfully used to treat 2 patients with recurrent Clostridium difficile infection (rCDI). Thus far, MET-2 has been studied in 14 human patients with rCDI. While the composition of MET-2 and MET-4 treatments are different, MET-4 contains several of the same bacteria present in MET-2.

ROMA LA-OPSCC-001 is a minimal risk feasibility study to evaluate the oral and intestinal microbiome using saliva, oropharyngeal swabs over tumor sites, stool and rectal swabs in patients with locoregionally-advanced oropharyngeal squamous cell carcinoma (LA-OPSCC) treated with chemoradiotherapy (CRT). This study involved analysis of samples from a prospective cohort of up to 30 patients diagnosed with LA-OPSCC treated with CRT. The study did not involve any therapeutic intervention. ROMA LA-OPSCC-001 is closed to accrual. A total of 181 samples have been collected. There was similarity in profiles between stool and rectal swab samples, and also between oropharyngeal swabs over the tumor site and saliva, but distinct by anatomical site, indicating that these sample types are able to resolve similarities by subject but distinguish anatomical compartments.

This data supports the study feasibility, compliance of sample acquisition and technical proficiency of characterizing the taxa composition at baseline and after CRT by using 4 methods of sample collection and suggest a potential treatment effect on both oral and intestinal microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written and voluntary informed consent.
2. Patient must be willing and able to provide:

   -Oropharyngeal swab, stool and blood specimen at protocol specified time points.
3. Age > 18 years, male or female.
4. Patient must be diagnosed with histologically confirmed squamous cell carcinoma of the oropharynx (soft palate, tonsils, base of tongue).
5. Patients must be eligible for curative-intent concurrent treatment with radiotherapy and chemotherapy.

Exclusion Criteria:

1. Any condition that, in the opinion of the Investigator, would interfere with patient safety, or evaluation of the collected specimen and interpretation of study result.
2. Subjects unable to swallow orally administered medications or any subjects with gastrointestinal disorders likely to interfere with absorption (e.g. bowel obstruction, short gut syndrome, blind loop syndrome, ileostomy etc). Subjects with colostomies may be enrolled.
3. Pregnant or planning to get pregnant in the next 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Toxicity defined by CTCAE v.5.0. | 1 year
  Safety and toxicity profile of MET-4 when administered concurrent to CRT.
Relative abundance of MET-4 associated bacterial strains in stool samples collected at week 4, end of CRT and 2-month follow-up timepoints. | 3 months
  Presence of MET-4 associated Operational taxonomic units (OTUs) in stool samples at specified timepoints.

SECONDARY OUTCOMES:
Bacterial composition and diversity between baseline, week 4, end of CRT and 2 month follow-up samples | 4 months
  DNA extraction from swabs/stool using Zymo Bacterial DNA Mini Prep, then 16S rRNA amplification and high throughput sequencing using Illumina Miseq to create an amplicon library from individual samples, then bioinformatic analysis, then shotgun metagenomics sequencing on an Illumina NextSeq, strain and species-specific qPCR for MET isolates and Nanostring nucleic acid detection using a custom array designed to quantitate MET-4 species will be performed in stool samples collected.
Bacterial composition and diversity of oral and stool samples in ROMA 1 (CRT alone) compared to ROMA 2 (CRT plus MET-4). | 4 months
  DNA extraction from swabs/stool using Zymo Bacterial DNA Mini Prep, then 16S rRNA amplification and high throughput sequencing using Illumina Miseq to create an amplicon library from individual samples, then bioinformatic analysis, then shotgun metagenomics sequencing on an Illumina NextSeq, strain and species-specific qPCR for MET isolates and Nanostring nucleic acid detection using a custom array designed to quantitate MET-4 species will be performed in stool samples collected.

OTHER OUTCOMES:
Correlation between blood immune profiling and changes in oral/intestinal microbiome in the context of CRT and MET-4 administration. | 1 year
  Immune profiling at specified timepoints.
Correlation between oral/intestinal microbiome and radiomics imaging analysis. | 1 year
  Tumor radiomic signatures before and after CRT.
Stool and serum metabolomic profiles before/after CRT and MET-4. | 1 year
  Metabolomics correlates at specified timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Spreafico, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No